CLINICAL TRIAL: NCT05534295
Title: Strokecopilot: A Precision Medicine Tool in the Stroke Emergency
Acronym: Strokecopilot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8589
Record Dates: First submitted 2022-09-02; First posted 2022-09-09 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cerebrovascular Accident (CVA)
Keywords: cerebrovascular accident (CVA); Ischemic stroke; thrombolysis channels; intravenous thrombolysis; mechanical thrombectomy
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ischemic stroke or cerebral infarction (CI) is an immediate emergency affecting approximately 100,000 - 150,000 patients each year in France and is managed in the neurovascular intensive care unit (NICU). Recanalization treatments can prevent disability, but patients must be carefully selected. Knowledge in this field is evolving rapidly, which tends to make management more complex and personalized. In addition, the permanence of thrombolysis channels involves neurologists of all expertise. Decision support tools are desirable to enable precision medicine in stroke. Strokecopilot is a web application developed by the principal investigator. Its algorithm contextualizes the patient in a set of evidence-based medicine references (recommendations and clinical trials) and gives the result of their cross-referencing to the user to indicate theoretical indications for intravenous thrombolysis and mechanical thrombectomy.

ELIGIBILITY:
Inclusion criteria:

- Adult patient (>18 years old) admitted to the thrombolysis unit of the University Hospital of Strasbourg from January 01, 2017 to December 31, 2021

Exclusion criteria:

- Subjects who have expressed their opposition to the use of their data for scientific research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient (>18 years old) admitted to the thrombolysis unit of the University Hospital of Strasbourg
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of thrombolysis data for the development of an algorithm to detect thrombolysis | Files analysed retrospectively from January 01, 2017 to December 31, 2021 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WOLFF, MD, PhD, Principal Investigator — Service : Unité Neurovasculaire - CHU de Strasbourg - France; Stanislas DEMUTH, MD, Principal Investigator — Service : Unité Neurovasculaire - CHU de Strasbourg - France
Locations (1):
- Service : Unité Neurovasculaire - CHU de Strasbourg - France, Strasbourg, France